CLINICAL TRIAL: NCT05985811
Title: Ketamine Analgesia Enhances Functional Quality and Mood in Chronic Pain Patients
Brief Title: Ketamine Enhances Analgesia and Mood in Chronic Pain Patients
Status: Recruiting | Type: Observational
Sponsor: Salem Anaesthesia Pain Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: SalemAnes2018 Ketamine Mood
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Mood Disorder; Opioid; Mood Insomnia
Keywords: Mood therapy
MeSH Terms: conditions — Mood Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Most chronic pain patients have mood disorders. The mood disorders may improve with better analgesia produced by Ketamine injections. A prospective study of patients undergoing interventional pain therapy using Ketamine injections. Pre-injection and post-injection patient data is collected. Pain is measured using numeric pain rating scale, and change in pain score by 2-points is considered significant. Sleep is measured using Likert sleep scale, and change in sleep score by 2-points is considered significant. Anxiety is measured using general anxiety disorder (GAD-7) scale, and change in anxiety score by 4-points is considered significant. Depression is measured using patient health questionnaire (PHQ-9), and change in depression score by 5-points is considered significant.

DETAILED DESCRIPTION:
Chronic pain is usually associated with psychological and mood disorders. Many chronic pain patients have various forms of mood abnormalities; and these mood issues may improve with better analgesia produced by Ketamine injections.

This is a prospective observational study of consenting adult patients who are undergoing interventional pain management. The patients undergo routine interventional pain therapy using Ketamine injections. Pre-injection and post-injection patient data is collected using validated tools. Data collection includes patients' age, psychiatric diagnosis, pain score, sleep score, anxiety score and depression score.

Pain score is measured using the numeric pain rating scale, and a change in the pain score by 2-points is considered significant. Sleep score is measured using the Likert sleep scale, and a change in the sleep score by 2-points is considered significant. Anxiety is measured using the general anxiety disorder (GAD-7) scale, and a change in the anxiety score by 4-points is considered significant. Depression is measured using the patient health questionnaire (PHQ-9) scale, and a change in the depression score by 5-points is considered significant.

Data is analyzed with IBM® SPSS® Statistics 25; using Student's t-test, ANOVA, Pearson Chi-square test, and regression analysis. P-value <0.05 is considered significant.

ELIGIBILITY:
Inclusion Criteria:

* adult chronic pain patients
* associated mood disorder
* good treatment compliance
* associated chronic insomnia
* regular ketamine pain therapy injection
* consent for clinical record quality assurance review

Exclusion Criteria:

* severe cognitive disorder
* inability to provide consent
* major neuropsychiatric disorder
* cannabis use
* stimulant use
* substance abuse
* poor treatment compliance
* lack of ketamine pain therapy injection

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult chronic pain clinic patients who have mood disorders; and undergoing routine regular ketamine injections for pain therapy.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-02-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain score, objective measurement using the validated Numeric Pain Rating scale | 12 weeks
  Pain score, using the Numeric Pain Rating scale of 0 to 10, low scores indicate less pain, high scores indicate worse pain

SECONDARY OUTCOMES:
Sleep quality score, objective measurement using the validated Likert sleep scale | 12 weeks
  Sleep quality score, using the Likert sleep scale of 0 to 10, low scores indicate poor sleep, high scores indicate better sleep

CONTACTS AND LOCATIONS:
Overall Officials: Olumuyiwa Bamgbade, MD,FRCPC, Principal Investigator — Salem Anaesthesia Pain Clinic
Locations (1):
- Salem Anaesthesia Pain Clinic, Surrey, British Columbia, Canada